CLINICAL TRIAL: NCT06686498
Title: Impact of a Recovery Model-based Intervention Targeting Adult Repeat Suicide Attempters: a Transformative Mixed Evaluation
Brief Title: Transformative Mixed Evaluation of a Suicide Attempt Recovery Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oriana Arellano Faúndez (Other)
Responsible Party: Sponsor-Investigator, Oriana Arellano Faúndez, Principal Investigator, Universidad Católica del Maule
Organization: Universidad Católica del Maule (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N°78/2024; N° 21221222. (Other: National Research and Development Agency (ANID))
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Suicidal Ideation; Suicidal Ideation and Behaviors
Keywords: recovery; reattempters suicide; evaluation; mixed method; intervention; adults
MeSH Terms: conditions — Suicidal Ideation; Behavior

STUDY DESIGN:
Intervention Model Description: In coherence with the recovery model and from a transformative paradigm, to meet the objectives, a mixed research study will be conducted, with a concurrent design constituted by two collection threads "QUAN (quantitative) and QUAL (qualitative)". This design is characterized by collecting, analyzing, and merging quantitative and qualitative data and results simultaneously, opting for one paradigm at the base rather than mixing paradigms.
  The longitudinal-type quantitative strand comprises a single-blind Randomized Clinical Trial (RCT) with two arms in parallel, in which two groups are compared: a waiting group that will function as a control group, which will receive its treatment as usual (TAU) called Group A. Furthermore, an experimental group called Group B, will receive both the usual treatment (TAU) and the IMR-ACS intervention. For ethical considerations, Group A will receive the
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual treatment (No Intervention): A waiting group that will function as a control group, which will receive its treatment as usual (TAU) called Group A. For ethical considerations, Group A will receive intervention once its impact has been proven through the present study
- Intervention and usual treatment (Experimental): An experimental group called Group B, will receive both the usual treatment (TAU) and the intervention.
  Interventions: Behavioral: Illness Management and Recovery adapted to suicidal behavior (IMR-ACS)

INTERVENTIONS:
Behavioral: Illness Management and Recovery adapted to suicidal behavior (IMR-ACS) — Illness Management and Recovery adapted to suicidal behavior (IMR-ACS) is a protocolized clinical intervention in a brief group format aimed at people at risk of suicide. Specifically, people who have had more than two attempts in their lifetime are called repeaters. For its construction, we relied on the Spanish version of the Illness Management and Recovery IMR, developed by the Spanish Nursing Association, adapted to the field of suicidal behavior, taking as a reference the model of personal recovery from suicide attempt proposed by Sokol et al.
  The goals of IMR-ACS are to 1) know the warning signs of a suicidal crisis, 2) implement strategies to manage the suicidal crisis, 3) foster social support among peers, 4) formulate goals for recovery from a suicidal crisis, and 5) seek help and make informed decisions in the event of a suicidal crisis.
  IMR-ACS is a complementary intervention to the usual treatments.
  Arms: Intervention and usual treatment

SUMMARY:
This study aims to evaluate the impact of a brief clinical group intervention based on the recovery model aimed at adult repeat suicide attempters attending an outpatient unit belonging to a public hospital in the Maule region, comparing two groups, one experimental and one wait group, considering indicators of clinical recovery (suicidal ideation, repetition of suicide attempt, functional disability, depressive symptoms), life satisfaction, social support, user satisfaction and personal recovery experiences lived by adult repeat suicide attempters.

DETAILED DESCRIPTION:
Suicide is a highly prevalent social and public health problem globally, nationally, and regionally. Globally, between 2000 and 2019, the suicide rate has decreased, except in the Americas, where rates increased by 17%. In Chile, according to World Bank data, the rate for the period 2000 to 2019 was nine deaths per 100,000 population, increasing to 10.3 after the COVID-19 pandemic. At the local level, there was a 51% increase in suicide attempts between 2019 and 2022. Additionally, self-inflicted injuries exhibited a 167% surge between 2018 and 2022, thereby elevating the risk of suicide, Despite this, suicide prevention interventions are characterized by being of an individual nature, based on risk and clinical indicators, and with an unproven impact, with even scarcer evidence on intervention models in suicide attempt repeaters. Although, a suicide attempt is the most critical predictor of lethal reattempts or death, especially in people presenting mood disorders.

Traditionally, both research and intervention on suicidal behavior have been approached mainly from the notion of risk, which has not brought, as in the Chilean case, favorable results in reducing suicide rates. This requires incorporating promotional, alternative, and complementary approaches that not only focus on reducing the variables that lead to suicide but also on the recovery of people after a suicidal episode. A positive life trajectory after a suicide attempt is extremely limited in research despite its advantage in helping to obtain favorable outcomes The recovery model implies a change in the view on mental health intervention, as it recognizes people's strengths and capabilities and transforms their role from that of the patient to that of the citizen. The model is closely related to social justice and places the person at the center.

In the field of suicidal behavior, adopting a recovery model constitutes a relevant strategy for suicide prevention, which does not imply leaving aside models focused on risk factors, but complementing it with an approach that takes into account the person in his or her family, social and cultural context.

Recovering after an attempt involves taking control of one's life and establishing a new daily life. It is a process that can be facilitated and constrained by a socio-structural context and can be referred both to clinical recovery, understood as a change in scores from a clinical to a non-clinical range on a series of measures capturing suicidal ideation and likelihood of suicide attempt, as to personal recovery, understood as a process of reconnecting with oneself while struggling with the death wish, which involves achieving a sense of agency, overcoming stigma, gaining social support, and developing social roles.

The present study aims to evaluate the impact of a recovery-based intervention considering indicators of clinical recovery (suicidal ideation, suicide attempt, functional disability), life satisfaction, user satisfaction, social support, and personal recovery experiences lived by adults' repeaters of suicide attempts, attended in an outpatient mental health center in the Maule region recognizing their socio-structural context.

Based on a transformative paradigm, the "QUAN + QUAL" concurrent mixed design integrates two data collection threads. A quantitative thread characterized by a single-blind randomized clinical trial with two parallel arms and a qualitative thread with a descriptive phenomenological design.

The proposed impact evaluation, by focusing on both clinical and personal recovery and the socio-structural context in which it is framed, allows us to address a notion of impact that recognizes the complex and processual nature of recovery for people with a history of suicide attempts.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age.
2. having made at least two suicide attempts in their lifetime,
3. presenting suicidal ideation (active or passive)
4. receiving individual outpatient treatment for a diagnosis of depression in a specialized mental health center, belonging to a Chilean Public Hospital, with a moderate-severe to severe level according to references from the clinical team

Exclusion Criteria:

1. to present dual pathology, active psychosis, cognitive or physical impairment, or other problems that impede the ability to understand the study procedures and give informed consent
2. to have participated in a group intervention related to mental health issues during the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of suicide attempts in the last month | From enrollment until 6 months after intervention is completed
  Report clinical team
Severity of Suicidal Ideation | From enrollment until 6 months after intervention is completed
  Columbia University Assessment of Suicidal Ideation Intensity Scale, C-SSRS Chile/Spanish 5.1 It includes six items with four Likert-type response options. Scoring: Minimum 0 points - Maximum 6 points. A higher score indicates greater severity of suicidal ideation.
Level of Functional Disability | From enrollment until 6 months after intervention is completed
  Questionnaire for the Assessment of Functional Disability self-administered version, WHODAS 2.0.
  The WHODAS 2.0 is a 12-item questionnaire that assesses six domains of functioning across physical and mental health disorders in clinical and non-clinical populations: cognition, mobility, self-care, getting along, life activities, and participation. Items are scored on a 5-point Likert scale ranging from 1 (None) to 5 (Extreme or cannot do) and are summed to create total and domain scores. Scores: Minimum 12 points - Maximum 60 points. A higher score indicates a higher level of total and domain disability.
Satisfaction with life | From enrollment until 6 months after intervention is completed
  Satisfaction with Life Scale. The SWLS, a measure of global cognitive judgments of life satisfaction, will be used to measure life satisfaction. Individuals provide a self-report response to five items on a 7-point Likert scale. Items are summed for a total score that can range from 5 to 35, with increasing scores indicating increased satisfaction with life. The SWLS has demonstrated good reliability and validity.
Social Support | From enrollment until 6 months after intervention is completed
  Perceived Social Support Scale, MOS. The scale consists of 19 items with a 5-point Likert-type response format. The first item measures the size of the social network, and the remaining items measure 4 dimensions of perceived social support: positive social interaction, affective, instrumental and emotional/informational support. Scores: Minimum 19 points - Maximum 60 points. A higher score indicates a higher level of social support overall and by dimension.
User satisfaction | From registration and at the end of the intervention
  Customer Satisfaction Questionnaire, CSQ-8. It includes eight items with four Likert-type response options. Scores: Minimum 8 points - Maximum 32 points. A higher score indicates a higher level of user satisfaction.
Depression | From enrollment until 6 months after intervention is completed
  Patient Health Questionnaire, PHQ9. The PHQ-9 is a screening scale that measures the presence and severity of depressive symptoms, and consists of 9 items with a 3-point Likert-type response format. Scores: Minimum 0 points - Maximum 27 points. A higher score indicates greater severity of depressive symptoms.
Socio-structural contextual/ | From enrollment until 6 months after intervention is completed
  Sociodemographic questionnaire: sex/gender, socioeconomic status, educational level, ethnicity, employment and housing status, etc. Variables measured ordinally, dichotomously, and nominally.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo I Méndez-Bustos, PhD, Study Director — Universidad Católica del Maule
Locations (1):
- Hospital Gral. Carlos Ibañez del Campo, Linares, Del Maule, Chile

IPD SHARING:
Plan to Share IPD: No
For ethical safeguards, the information that will be shared will be unaggregated and anonymized.

REFERENCES:
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Mueser, K. (2013). Illness Management and Recovery. SAMSHA´S GAINS Center for Behavioral Health and Justice Transformation https://www.usf.edu/cbcs/mhlp/tac/documents/behavioral-healthcare/samh/illness-management-and-recovery.pdf
- [Background] Mueser KT, Meyer PS, Penn DL, Clancy R, Clancy DM, Salyers MP. The Illness Management and Recovery program: rationale, development, and preliminary findings. Schizophr Bull. 2006 Oct;32 Suppl 1(Suppl 1):S32-43. doi: 10.1093/schbul/sbl022. Epub 2006 Aug 9. PMID 16899534
- [Background] Mueser KT, Corrigan PW, Hilton DW, Tanzman B, Schaub A, Gingerich S, Essock SM, Tarrier N, Morey B, Vogel-Scibilia S, Herz MI. Illness management and recovery: a review of the research. Psychiatr Serv. 2002 Oct;53(10):1272-84. doi: 10.1176/appi.ps.53.10.1272. PMID 12364675
- [Background] Mertens, D. M. (2021). Transformative research methods to increase social impact for vulnerable groups and cultural minorities. International Journal of Qualitative Methods, 20. https://doi.org/10.1177/16094069211051563
- [Background] Asociación Española de Enfermería de Salud Mental (2020). Manejo y Recuperación de un problema de salud mental grave (IMR). Adaptación al español de Substance Abuse and Mental Health Services Administration (2009). Illness Management and Recovery: Practitioner Guides and Handouts. HHS Pub. No. SMA-09-4462, Rockville, MD: Center for Mental Health Services, Substance Abuse and Mental Health Services Administration, U.S. Department of Health and Human Services.
- [Background] Ropaj E, Haddock G, Pratt D. Developing a consensus of recovery from suicidal ideations and behaviours: A Delphi study with experts by experience. PLoS One. 2023 Sep 20;18(9):e0291377. doi: 10.1371/journal.pone.0291377. eCollection 2023. PMID 37729121
- [Background] Karadzhov D. Personal recovery and socio-structural disadvantage: A critical conceptual review. Health (London). 2023 Mar;27(2):201-225. doi: 10.1177/13634593211014250. Epub 2021 May 7. PMID 33962518
- [Background] Sokol Y, Levin C, Linzer M, Rosensweig C, Hubner S, Gromatsky M, Walsh S, Dixon L, Goodman M. Theoretical model of recovery following a suicidal episode (COURAGE): scoping review and narrative synthesis. BJPsych Open. 2022 Nov 17;8(6):e200. doi: 10.1192/bjo.2022.599. PMID 36384945
- [Background] Espeland K, Loa Knizek B, Hjelmeland H. Lifesaving turning points: First-person accounts of recovery after suicide attempt(s). Death Stud. 2023;47(5):550-558. doi: 10.1080/07481187.2022.2108941. Epub 2022 Aug 8. PMID 35939504